CLINICAL TRIAL: NCT04102943
Title: Single Center, Randomized, Open-label, Phase IV Study to Evaluate the Pharmacokinetics and Tolerability of Tacrolimus Tablet(TacroBell) in Kidney Transplant Recipients.
Brief Title: Study to Evaluate the Pharmacokinetics and Tolerability of Tacrolimus in Kidney Transplant Recipients.
Acronym: PK-TACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211KT17009
Record Dates: First submitted 2019-08-28; First posted 2019-09-25 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus1 (Experimental): Tacrolimus tablet Orally, twice a day in the morning and night After first dose 0.1mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 7~12ng/ml for 0 to 3months and then at 5~8ng/ml for 3 to 6months of study treatment.
  Interventions: Drug: tacrolimus tablet
- Tacrolimus2 (Active Comparator): Tacrolimus Cap Orally, twice a day in the morning and night After first dose 0.1mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 7~12ng/ml for 0 to 3months and then at 5~8ng/ml for 3 to 6months of study treatment.
  Interventions: Drug: tacrolimus capsules

INTERVENTIONS:
Drug: tacrolimus tablet — * Orally, twice a day in the morning and night
  * After first dose 0.1mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 7~12ng/ml for 0 to 3months and then at 5~8ng/ml for 3 to 6months of study treatment.
  Other Names: tacrobell tablet
  Arms: Tacrolimus1
Drug: tacrolimus capsules — * Orally, twice a day in the morning and night
  * After first dose 0.1mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 7~12ng/ml for 0 to 3months and then at 5~8ng/ml for 3 to 6months of study treatment.
  Other Names: prograf capsules
  Arms: Tacrolimus2

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and tolerability of Tacrolimus tablet(TacroBell) in kidney transplant recipients.

DETAILED DESCRIPTION:
This study is a Single center, randomized, open-label, Phase IV study to evaluate the pharmacokinetics and tolerability of Tacrolimus tablet(TacroBell) administration for 24 Weeks in patients after renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years old(male or female)
* Patients who are planning to receive a kidney from a deceased or a living non-related/related donor
* Agreement with written informed consent

Exclusion Criteria:

* Previously received organs other than kidneys or who are planed to be transplanted simultaneously
* Diagnosed with cancer in the last five years [Patients, however, who have recovered from skin cancer (squamous cell/basal cell carcinoma) or thyroid cancer can be enrolled.]
* Patients or donors who have positive HIV test result
* Inadequate for registration under the judgment of the investigator due to severe gastrointestinal disorders
* Severe systemic infection requiring treatment
* Prior to the kidney transplantation

  * Treatment with active liver disease or Liver function test(T-bilirubin, Aspartate transaminase(AST), Alanine transaminase(ALT))is over 3 times than upper normal limit
  * White Blood Cell(WBC) <2.5 x10^3/μL, or platelet <75 x10^3/μL
* Pregnant women or nursing mothers
* Fertile women who not practice contraception with appropriate methods
* Participated in other trial within 4 weeks
* In investigator's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-08-28 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Cmax (Maximum concentration of drug in serum) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours)
  Measurement of TDM of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
AUCt (Area under the plasma concentration-time curve from time zero to time t) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours)
  Measurement of TDM of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules

SECONDARY OUTCOMES:
Tmax (Time of peak concentration) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
AUC∞ (Area under the plasma concentration-time curve from time zero to infinity) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Cmax (Maximum concentration of drug in serum) | At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
AUCt (Area under the plasma concentration-time curve from time zero to time t) | At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of TDM of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Tmax (Time of peak concentration) | At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
AUC∞ (Area under the plasma concentration-time curve from time zero to infinity) | At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of TDM of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Dose normalized Cmax(Maximum concentration of drug in serum) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours), At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Dose normalized AUCt(Area under the plasma concentration-time curve from time zero to time t) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours), At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Dose normalized Tmax(Time of peak concentration) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours), At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules
Dose normalized AUC∞(Area under the plasma concentration-time curve from time zero to infinity) | At 2weeks predose(0hour)and dose(0.5,1,1.5,2,3,4,8,12hours), At 24weeks predose(0hour)and dose(0.5,1,1.5,2,3,4hours)
  Measurement of therapeutic drug concentration monitoring(TDM) of tacrolimus after administration of tacrolimus tablets or tacrolimus capsules

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea